CLINICAL TRIAL: NCT05027802
Title: Rollover Study; Multicentre, Phase III, Open-label Study to Further Evaluate the Safety and Efficacy of Palovarotene Capsules in Male and Female Participants Aged ≥14 Years With Fibrodysplasia Ossificans Progressiva (FOP) Who Have Completed Study PVO-1A-301 or PVO-1A-202/PVO-1A-204 and May Benefit From Palovarotene Therapy.
Brief Title: A Rollover Study to Further Evaluate the Safety and Efficacy of Palovarotene Capsules in Male and Female Participants Aged ≥14 Years With Fibrodysplasia Ossificans Progressiva (FOP) Who Have Completed the Relevant Parent Studies.
Acronym: PIVOINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-60120-452; 2021-002244-70 (EudraCT Number)
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Fibrodysplasia Ossificans Progressiva (FOP)
MeSH Terms: conditions — Myositis Ossificans | interventions — Palovarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Palovarotene Chronic/Flare-Up Regimen (Experimental): Chronic treatment: participants will receive 5 mg palovarotene or the dose received during participation in the parent study at the time of transition to Study CLIN-60120-452 or prior to interrupting/stopping palovarotene treatment.
  Flare-up treatment: at the time of a flare-up (or substantial high-risk traumatic event likely to lead to a flare-up) participants will receive 20 mg palovarotene for 28 days, followed by 10 mg palovarotene for 56 days.
  Interventions: Drug: Palovarotene

INTERVENTIONS:
Drug: Palovarotene — Palovarotene will be taken orally once daily at approximately the same time each day.

SUMMARY:
The main objective of this study is to further evaluate the safety and efficacy of palovarotene in adult and paediatric participants with FOP.

The aim of the study is also to ensure treatment continuity to participants who have completed one of the parent studies (Study PVO-1A-301, Study PVO-1A-202 and Study PVO-1A-204) and who, in the investigator's judgement, may benefit from palovarotene therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed the EOS or End of Treatment Visit of Study PVO-1A-301 or PVO-1A-202 (PVO-1A-202 Parts C and D correspond to Study PVO-1A-204 in France) and did not previously withdraw consent from any of the parent studies to be eligible for Study CLIN-60120-452.
* Participant must be ≥14 years of age (aligned with the age of treated participants in the ongoing parent studies PVO-1A-301 and PVO-1A-202/PVO-1A-204) and qualify as 100% skeletally mature (if <18 years, based on assessments carried out at parent EOS Visit; if ≥18 years, automatically considered 100% skeletally mature) or have reached final adult height based on investigator's assessment, at the time the Study CLIN- 60120-452 informed consent is signed.

Exclusion Criteria:

* History of allergy or hypersensitivity to retinoids, gelatin, lactose (note that lactose intolerance is not exclusionary) or palovarotene, or unresponsiveness to prior treatment with palovarotene.
* Uncontrolled cardiovascular, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, ophthalmologic, immunologic, psychiatric, or other significant disease.
* Symptomatic vertebral fracture.
* Intercurrent known or suspected non-healed fracture at any location;
* Any other medical condition/clinically significant abnormalities that would expose the participant to undue risk or interfere with study assessments.
* Amylase or lipase >2× above the upper limit of normal (ULN) or with a history of chronic pancreatitis.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5× ULN.
* Fasting triglycerides >400 mg/dL with or without therapy.
* Suicidal ideation (type 4 or 5) or any suicidal behaviour at the Inclusion Visit as defined by the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Current use of vitamin A or beta carotene, multivitamins containing vitamin A or beta carotene, or herbal preparations, fish oil, and unable or unwilling to discontinue use of these products during palovarotene treatment.
* Exposure to synthetic oral retinoids other than palovarotene within 4 weeks of the Inclusion Visit.
* Concurrent treatment with tetracycline or any tetracycline derivatives due to the potential increased risk of pseudotumor cerebri.
* Use of concomitant medications that are strong inhibitors or inducers of cytochrome P450 (CYP450) 3A4 activity; or kinase inhibitors such as imatinib.
* Palovarotene is reimbursed in the country where the study is being conducted.
* Any reason that, in the opinion of the investigator, would lead to the inability of the participant and/or family to comply with the protocol.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (13):
- United States (4):
  - University of California San Francisco (UCSF), San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of Philidelphia, Philadelphia, Pennsylvania
  - The Perelman School of Medicine - The University of Pennsylvania, Philadelphia, Pennsylvania
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Royal North Shore Hospital, Saint Leonards, New South Wales, Australia
- Hospital Israelita Albert Einstein, Morumbi, São Paulo, Brazil
- Toronto General Hospital, Toronto, Canada
- Groupe Hospitalier Necker Enfants Malades, Paris, France
- Istituto Giannina Gaslini, Genoa, Italy
- Hospital Universitario Ramon y Cajal, Colmenar Viejo, Spain
- Norrlands Universitetssjukhus, Umeå, Sweden
- Royal National Orthopaedic Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2025/06/11113724/CLIN-60120-452_Lay-Summary_Final_23May2025.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-arm, rollover, multicenter, Phase III, open-label study was conducted at 12 investigational sites in 9 countries from 14-Mar-2022 to 30-Nov-2024 in participants >=14 years with fibrodysplasia ossificans progressiva (FOP) who had completed parent study PVO-1A-301 (NCT03312634) or PVO-1A-202 (NCT02279095)/PVO-1A-204 (NCT02979769) and continued to benefit from palovarotene therapy. A total of 61 participants were enrolled in the study of which 59 received treatment.
Pre-assignment Details: This study consisted of an Inclusion visit which included signing of informed consent form (Day 1), a continuous dosing treatment period (including a follow-up visit every 6 months), and an end of study/early withdrawal visit. Participants were eligible for the study whether they received chronic or flare-up treatment in the parent study at the time of transition.
Groups:
- Palovarotene: Participants continued to receive palovarotene 5 milligram (mg) orally once daily until it was reimbursed in the country where the study was being conducted or another access program became available or until the study end date, whichever occurred first, up to approximately 32 months.
  In case of flare-up symptoms or substantial high risk traumatic events (likely to lead to a flare-up), participants received palovarotene 20 mg orally once daily for 4 weeks followed by 10 mg orally once daily for 8 weeks for a total of 12 weeks even if symptoms resolved earlier.
Period: Overall Study
Arm/Group | Palovarotene
Started (Enrolled) | 61
Received Treatment | 59
Completed | 38
Not Completed | 23
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 18
Not completed — Death | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS)/safety set included all participants who received at least 1 dose of palovarotene in this study.
Groups:
- Palovarotene: Participants continued to receive palovarotene 5 mg orally once daily until it was reimbursed in the country where the study was being conducted or another access program became available or until the study end date, whichever occurred first, up to approximately 32 months.
  In case of flare-up symptoms or substantial high risk traumatic events (likely to lead to a flare-up), participants received palovarotene 20 mg orally once daily for 4 weeks followed by 10 mg orally once daily for 8 weeks for a total of 12 weeks even if symptoms resolved earlier.
Arm/Group | Palovarotene
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38
  Black or African American | 0
  Asian | 3
  Other | 1
  Multiple | 2
  Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Treatment-emergent Adverse Events (TEAEs), Serious and Non-serious Treatment-emergent Adverse Events and Serious and Non-serious Treatment-related Treatment-emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or significant medical event. A TEAE was defined as any AE that occurred after signing the informed consent form of this study or an ongoing AE from the parent study with a worsening in severity or relationship to the study treatment following transition to this study.
Time Frame: From signing the informed consent form (Day 1) up to 30 days post last dose, approximately 32 months
Population: The FAS/safety set included all participants who received at least 1 dose of palovarotene in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 59
Participants
  All TEAEs | 54
  Serious TEAEs | 9
  Non-serious TEAEs | 53
  Serious treatment-related TEAEs | 1
  Non-serious treatment-related TEAEs | 38

2. Secondary Outcome: Change From the Inclusion Visit in Cumulative Analogue Joint Involvement Scale (CAJIS) Total Score at Months 6, 12, 18, 24 and 30
Description: The CAJIS is an objective measure of joint movement completed by the investigator to document total joint involvement. This scale assesses functional disability by categorizing range of motion across 12 joints (both right and left shoulder, elbow, wrist, hip, knee and ankle joints) and 3 body regions (cervical spine, thoracic/lumbar spine and jaw), with each joint/region assessed as: 0=normal (<10% deficit); 1=partially impaired (10% to 90% deficit) and 2=functionally ankylosed (>90% deficit). The CAJIS total score is calculated as the sum of the scores of all joints/regions and ranges from 0 (no involvement) to 30 (maximally involved). Higher score indicated worse outcome. The Inclusion Visit was the first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: The FAS/safety set included all participants who received at least 1 dose of palovarotene in this study. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Palovarotene
Number analyzed (Participants) | 53
score on a scale
  Month 6: number analyzed (Participants) | 52
  Month 6 | 0.6 (1.3)
  Month 12 | 1.1 (2.0)
  Month 18: number analyzed (Participants) | 45
  Month 18 | 1.5 (2.3)
  Month 24: number analyzed (Participants) | 25
  Month 24 | 1.5 (2.6)
  Month 30: number analyzed (Participants) | 8
  Month 30 | 2.0 (4.7)

3. Secondary Outcome: Change From the Inclusion Visit in the Use of Assistive Devices and Adaptations (Aids) for Daily Living at Months 6, 12, 18, 24 and 30
Description: The use of assistive devices and adaptations (aids) for daily living was collected using the FOP assistive devices assessment at each visit. Assistive devices and adaptations include mobility aids, eating tools, personal care tools, bathroom aids and devices, bedroom aids and devices, home adaptions, work environment adaptions, technology adaptions, sports and recreation adaptions, school adaptions and medical therapies for daily living. The mean of total number of assistive devices and adaptations for daily living being used is presented. The Inclusion Visit was the first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of aids
Arm/Group | Palovarotene
Number analyzed (Participants) | 53
number of aids
  Month 6 | -0.7 (3.4)
  Month 12: number analyzed (Participants) | 51
  Month 12 | 1.1 (4.7)
  Month 18: number analyzed (Participants) | 46
  Month 18 | 1.4 (5.7)
  Month 24: number analyzed (Participants) | 23
  Month 24 | 1.2 (5.1)
  Month 30: number analyzed (Participants) | 6
  Month 30 | 2.8 (7.4)

4. Secondary Outcome: Change From the Inclusion Visit in Percentage of Worst Score Using the Adult Form of the Fibrodysplasia Ossificans Progressiva Physical Function Questionnaire (FOP-PFQ) at Months 6, 12, 18, 24 and 30
Description: The FOP-PFQ is a disease-specific patient-reported outcome measure of physical impairment; includes 28 questions related to activities of daily living and physical performance scored on a scale of 1 to 5 with lower scores indicating that participant has more difficulty completing those tasks. Total score, upper extremities subscore and mobility subscore is calculated as follows: total score: sum of the scores from each question (range 28 to 140); upper extremities subscore: sum of the scores from 15 questions (questions 1-12, 14, 25 and 26; range 15 to 75); mobility subscore: the sum of the scores from 13 questions (questions 13, 15-24, 27 and 28; range 13 to 65). The scores were transformed to reflect a percentage of worst score which ranged from 0% to 100% with 0% indicating the best possible function and 100% (higher score) indicating the worst possible function. Mean is presented. Inclusion Visit was first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | Palovarotene
Number analyzed (Participants) | 54
percentage of score
  Month 6: total score | 0.74 (6.37)
  Month 12: total score: number analyzed (Participants) | 52
  Month 12: total score | 2.39 (10.21)
  Month 18: total score: number analyzed (Participants) | 47
  Month 18: total score | 4.77 (12.39)
  Month 24: total score: number analyzed (Participants) | 25
  Month 24: total score | 7.80 (15.15)
  Month 30: total score: number analyzed (Participants) | 9
  Month 30: total score | 13.79 (21.98)
  Month 6: upper extremities subscore | 0.70 (6.87)
  Month 12: upper extremities subscore: number analyzed (Participants) | 52
  Month 12: upper extremities subscore | 1.12 (8.52)
  Month 18: upper extremities subscore: number analyzed (Participants) | 47
  Month 18: upper extremities subscore | 3.24 (11.28)
  Month 24: upper extremities subscore: number analyzed (Participants) | 25
  Month 24: upper extremities subscore | 5.54 (12.42)
  Month 30: upper extremities subscore: number analyzed (Participants) | 9
  Month 30: upper extremities subscore | 8.15 (11.50)
  Month 6: mobility subscore | 0.74 (9.15)
  Month 12: mobility subscore: number analyzed (Participants) | 52
  Month 12: mobility subscore | 3.90 (14.98)
  Month 18: mobility subscore: number analyzed (Participants) | 47
  Month 18: mobility subscore | 6.53 (17.45)
  Month 24: mobility subscore: number analyzed (Participants) | 25
  Month 24: mobility subscore | 10.38 (23.08)
  Month 30: mobility subscore: number analyzed (Participants) | 9
  Month 30: mobility subscore | 20.30 (36.44)

5. Secondary Outcome: Annualized Rate of Healthcare Utilization (HU) in Participants With Fibrodysplasia Ossificans Progressiva
Description: Annualized HU rate was defined as the (number of HU during the study/duration of participant participation in the study in days) * 365.25. Annualized rate for total health care services utilized is presented.
Time Frame: Up to approximately 32 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: HU per participant year
Arm/Group | Palovarotene
Number analyzed (Participants) | 55
HU per participant year | 21.7 (31.4)

6. Secondary Outcome: Change From the Inclusion Visit in Percent Predicted Forced Vital Capacity (FVC) at Months 6, 12, 18, 24 and 30
Description: Lung function parameters including FVC were obtained by spirometry. The Inclusion Visit was the first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Palovarotene
Number analyzed (Participants) | 38
percent predicted FVC
  Month 6: number analyzed (Participants) | 17
  Month 6 | 1.2 (5.5)
  Month 12 | -0.7 (6.8)
  Month 18: number analyzed (Participants) | 16
  Month 18 | -3.9 (9.8)
  Month 24: number analyzed (Participants) | 15
  Month 24 | -1.6 (5.8)
  Month 30: number analyzed (Participants) | 4
  Month 30 | -2.8 (3.8)

7. Secondary Outcome: Change From the Inclusion Visit in Percent Predicted Forced Expiratory Volume in One Second (FEV1) at Months 6, 12, 18, 24 and 30
Description: Lung function parameters including FEV1 were obtained by spirometry. The Inclusion Visit was the first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Palovarotene
Number analyzed (Participants) | 38
percent predicted FEV1
  Month 6: number analyzed (Participants) | 17
  Month 6 | 1.8 (5.9)
  Month 12 | -3.1 (9.6)
  Month 18: number analyzed (Participants) | 16
  Month 18 | -5.3 (11.8)
  Month 24: number analyzed (Participants) | 15
  Month 24 | -3.8 (6.6)
  Month 30: number analyzed (Participants) | 4
  Month 30 | -10.0 (11.1)

8. Secondary Outcome: Change From the Inclusion Visit in Predicted FEV1/FVC Ratio at Months 6, 12, 18, 24 and 30
Description: The ratio of FEV1 to FVC was calculated. Lung function parameters were obtained by spirometry. The Inclusion Visit was the first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palovarotene
Number analyzed (Participants) | 38
ratio
  Month 6: number analyzed (Participants) | 17
  Month 6 | 0.0163 (0.0574)
  Month 12 | -0.0323 (0.1358)
  Month 18: number analyzed (Participants) | 16
  Month 18 | -0.0137 (0.0888)
  Month 24: number analyzed (Participants) | 15
  Month 24 | -0.0365 (0.0994)
  Month 30: number analyzed (Participants) | 4
  Month 30 | -0.1268 (0.1564)

9. Secondary Outcome: Change From the Inclusion Visit in Percent Predicted Diffusion Capacity of the Lung for Carbon Monoxide (DLCO) at Months 6, 12, 18, 24 and 30
Description: The DLCO test provides information on the efficiency of gas transfer from alveolar air into the bloodstream. The Inclusion Visit was the first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted DLCO
Arm/Group | Palovarotene
Number analyzed (Participants) | 36
percent predicted DLCO
  Month 6: number analyzed (Participants) | 14
  Month 6 | -1.5 (7.9)
  Month 12 | -5.3 (12.6)
  Month 18: number analyzed (Participants) | 14
  Month 18 | -4.4 (16.5)
  Month 24: number analyzed (Participants) | 14
  Month 24 | -4.8 (11.4)
  Month 30: number analyzed (Participants) | 3
  Month 30 | -20.0 (20.3)

10. Secondary Outcome: Change From the Inclusion Visit in Physical and Mental Function Using Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale at Months 6, 12, 18, 24 and 30
Description: The PROMIS Global Health Scale is a patient-reported outcome measure of physical and mental function. The adult form (developed for participants >=15 years old) was used for all participants,consists of 10 questions from which 2 scores are calculated: global physical health score (GPH) and global mental health (GMH) score, each ranging from 4 (worse health) to 20 (better health). GPH score:sum of scores from Questions 3, 6, 7 and 8 and GMH score:sum of scores from Questions 2, 4, 5 and 10.These scores were converted to a T-score whose distributions were standardized such that value of 50 represented average (mean) for general population and increments of +/- 10 points represented +/- 1 standard deviation away from the norm.Higher T-scores indicated better physical/mental health. A T-score <50 indicated worse health than general population, while a T-score >50 indicated better health. Inclusion Visit was first study visit (Day 1) and first administration of palovarotene in this study.
Time Frame: Inclusion Visit (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Palovarotene
Number analyzed (Participants) | 54
T-score
  Month 6: GPH | -0.6 (4.4)
  Month 12: GPH: number analyzed (Participants) | 53
  Month 12: GPH | -1.7 (5.0)
  Month 18: GPH: number analyzed (Participants) | 48
  Month 18: GPH | -2.9 (5.0)
  Month 24: GPH: number analyzed (Participants) | 24
  Month 24: GPH | -1.9 (5.8)
  Month 30: GPH: number analyzed (Participants) | 8
  Month 30: GPH | -3.9 (7.0)
  Month 6: GMH | -1.0 (4.8)
  Month 12: GMH: number analyzed (Participants) | 53
  Month 12: GMH | -1.5 (6.3)
  Month 18: GMH: number analyzed (Participants) | 48
  Month 18: GMH | -2.3 (6.9)
  Month 24: GMH: number analyzed (Participants) | 24
  Month 24: GMH | -2.2 (6.0)
  Month 30: GMH: number analyzed (Participants) | 8
  Month 30: GMH | -5.7 (5.1)

11. Secondary Outcome: Number of Participants With Flare-ups and Flare-up Outcomes
Description: Number of participants with at least 1 flare-up and intercurrent flare-ups since last visit is presented. Intercurrent flare-ups were defined as a new flare-up or marked worsening of the original flare up at any time during a flare-up-based treatment cycle. Outcome of flare-ups resulting in movement restriction and bone formations in participants is presented. Movement restriction includes categories like better, same, slightly worse, moderately worse and severely worse movement than before.
Time Frame: Months 6, 12, 18 and 24
Population: The FAS/safety set included all participants who received at least 1 dose of palovarotene in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 59
Participants
  Month 6: at least 1 flare up since last visit | 27
  Month 12: at least 1 flare up since last visit | 26
  Month 18: at least 1 flare up since last visit | 15
  Month 24: at least 1 flare up since last visit | 4
  Month 6: intercurrent flare-ups since last visit | 7
  Month 12: intercurrent flare-ups since last visit | 4
  Month 18: intercurrent flare-ups since last visit | 4
  Month 24: intercurrent flare-ups since last visit | 0
  Month 6: better movement | 0
  Month 6: same movement | 22
  Month 6: slightly worse movement | 7
  Month 6: moderately worse movement | 5
  Month 6: severely worse movement | 1
  Month 12: better movement | 1
  Month 12: same movement | 17
  Month 12: slightly worse movement | 10
  Month 12: moderately worse movement | 5
  Month 12: severely worse movement | 0
  Month 18: better movement | 0
  Month 18: same movement | 7
  Month 18: slightly worse movement | 7
  Month 18: moderately worse movement | 1
  Month 18: severely worse movement | 1
  Month 24: better movement | 0
  Month 24: same movement | 1
  Month 24: slightly worse movement | 3
  Month 24: moderately worse movement | 0
  Month 24: severely worse movement | 1
  Month 6: bone formation | 5
  Month 12: bone formation | 5
  Month 18: bone formation | 1
  Month 24: bone formation | 0

12. Secondary Outcome: Number of Participants With Flare-ups by Body Location
Description: Number of participants with flare-ups by body locations including shoulder, elbow, hip, knee, ankle or foot, back, jaw and submandibular area and other (includes all other locations than mentioned) is presented.
Time Frame: Months 6, 12, 18 and 24
Population: The FAS/safety set included all participants who received at least 1 dose of palovarotene in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 59
Participants
  Month 6: shoulder | 8
  Month 6: elbow | 3
  Month 6: hip | 5
  Month 6: knee | 5
  Month 6: ankle or foot | 3
  Month 6: back | 4
  Month 6: jaw and submandibular area | 4
  Month 6: other | 14
  Month 12: shoulder | 4
  Month 12: elbow | 2
  Month 12: hip | 5
  Month 12: knee | 3
  Month 12: ankle or foot | 5
  Month 12: back | 2
  Month 12: jaw and submandibular area | 3
  Month 12: other | 12
  Month 18: shoulder | 4
  Month 18: elbow | 1
  Month 18: hip | 3
  Month 18: knee | 2
  Month 18: ankle or foot | 2
  Month 18: back | 1
  Month 18: jaw and submandibular area | 0
  Month 18: other | 8
  Month 24: shoulder | 1
  Month 24: elbow | 0
  Month 24: hip | 0
  Month 24: knee | 1
  Month 24: ankle or foot | 1
  Month 24: back | 0
  Month 24: jaw and submandibular area | 0
  Month 24: other | 2

13. Secondary Outcome: Duration of Flare-up at Months 6, 12, 18 and 24
Description: Duration of flare-up was defined as (date of end of flare-up - date of start of flare-up + 1).
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palovarotene
Number analyzed (Participants) | 27
days
  Month 6 | 130.7 (153.3)
  Month 12: number analyzed (Participants) | 26
  Month 12 | 121.7 (102.7)
  Month 18: number analyzed (Participants) | 15
  Month 18 | 72.4 (42.6)
  Month 24: number analyzed (Participants) | 4
  Month 24 | 72.3 (53.9)

14. Secondary Outcome: Percentage of Participants With Extra Bone Growth at Months 6, 12, 18 and 24
Description: Percentage of participants with at least 1 extra bone growth associated or not with a flare-up since last visit is presented.
Time Frame: Months 6, 12, 18 and 24
Population: The FAS/safety set included all participants who received at least 1 dose of palovarotene in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 59
percentage of participants
  Month 6: associated | 8.5
  Month 6: not associated | 3.4
  Month 12: associated | 8.5
  Month 12: not associated | 8.5
  Month 18: associated | 1.7
  Month 18: not associated | 3.4
  Month 24: associated | 0
  Month 24: not associated | 3.4

ADVERSE EVENTS:
Time Frame: Adverse events and deaths were collected from signing the informed consent form (Day 1) up to 30 days post last dose, approximately 32 months
Description: The FAS/safety set included all participants who received at least 1 dose of palovarotene in this study.
Arm/Group | Palovarotene
All-Cause Mortality (participants affected / at risk) | 2/59
Serious Adverse Events (participants affected / at risk) | 9/59
Other Adverse Events (participants affected / at risk) | 45/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene (N=59)
Pneumonia (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Callus formation delayed (Musculoskeletal and connective tissue disorders) | 1 (2)
Lymphoedema (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene (N=59)
COVID-19 (Infections and infestations) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Localised infection (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (5)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 10 (12)
Skin abrasion (Injury, poisoning and procedural complications) | 7 (8)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 4 (6)
Oedema peripheral (General disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Lip dry (Gastrointestinal disorders) | 4 (4)
Lung diffusion disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Lymphoedema (Vascular disorders) | 5 (5)
Drug hypersensitivity (Immune system disorders) | 5 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT05027802/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT05027802/SAP_001.pdf